## Statistical analysis plan

**Title of the study**: Split-in-situ Resection With Radio-frequency Ablation Instead of Liver Partition on the First Stage (RALPPS) in Patients With Hilar and Intrahepatic Cholangiocarcinoma

**Unic Protocol ID:** MCNC 09/2017

**Date:** October 24, 2017

## Statistical analysis

The propensity score matching (PSM) method was used to overcome heterogeneity of retrospectively collected data in compared groups. Nearestneighbor algorithm with 1:1 match ratio using a 0.2 caliper was applied. Matching for stage 1 included following factors: maximum total bilirubin level, duration of jaundice and acute cholangitis presence. PSM model for stage 2 enrolled FLR volume after portal vein occlusion (first stage). Continuous data presented as median values were compared using Mann Whitney U test before and after PSM. The Two-tailed Fisher's Exact test was used for comparing categorical variables before and after PSM. A p-value of less than 0.05 was considered statistically significant. SPSS version 23.0 (IBM SPSS, Inc., Chicago, IL) software package was applied for data analysis.

Mikhail Efanov, MD, PhD, Head of the HepatoPancreatoBiliary Surgery Department, Moscow Clinical Scientific Center +7(916) 105-88-30 www.mknc.ru